CLINICAL TRIAL: NCT01716338
Title: Glyburide Healthy Volunteer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-15112.b; NCT01157637 (obsolete NCT alias)
Record Dates: First submitted 2012-10-12; First posted 2012-10-29 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Volunteers
Keywords: glyburide; glybenclamide; hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glyburide; Sugars; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glyburide (Active Comparator): 1.5 mg (lowest dose) by mouth every day with breakfast for 7 days
  Interventions: Drug: Glyburide
- Sugar Pill (Capsule) (Placebo Comparator): Matching placebo capsule by mouth every day with breakfast for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glyburide
  Other Names: Micronase; Glybencamide
  Arms: Glyburide
Drug: Placebo
  Other Names: Sugar Pill (capsule)
  Arms: Sugar Pill (Capsule)

SUMMARY:
Glyburide is a medication that has been safely used for several decades to treat non-insulin dependent diabetes. This pilot study seeks to evaluate whether glyburide, administered at the lowest dose (1.5 mg/dL daily) to healthy (non-diabetic) subjects is safe both physically and cognitively. The investigators are hopeful that the results of this study will provide the necessary foundation to evaluate this medication's use on a larger scale to determine the feasibility of using glyburide in soldiers either prophylactically or for the treatment of brain injury.

DETAILED DESCRIPTION:
This study is a placebo controlled (2:1 drug vs. placebo), randomized clinical trial of 21 healthy, non-diabetic volunteers receiving daily doses of oral glyburide (1.5 mg) vs. placebo while under careful medical monitoring in an inpatient Clinical Research Unit (CRU)within the Center for Applied Research Sciences (CARS) at the Washington University in St. Louis Medical Center for a duration of 7 days and nights (24 hours per day). Interested subjects who call for more information about the study will be scheduled for a screening visit. Subjects will participate first in an informed consent process, and those wishing to take part will be asked to undergo a comprehensive interview detailing their past medical history and formal physical examination (which includes laboratory tests of the urine and blood). If a subject is deemed appropriate by the team, he/she will be asked to perform an exercise test (treadmill for 30 minutes) and will have an Electrocardiogram (ECG) completed to further determine eligibility. Individuals who do not meet inclusion criteria based on screening activities will be notified immediately that they are not eligible. Volunteers meeting all eligibility criteria will be scheduled for the week long in-patient evaluation.

Each subject will undergo a battery of physical, cognitive, and laboratory tests in addition to receiving oral glyburide or placebo each day for one week.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between the ages of 18 and 40.
* Have a Body Mass Index (BMI) between 18-30.
* Normal screening physical examination (non-pregnant as confirmed by serum Beta HcG,non-diabetic as confirmed by normal Hgb A-1C, normal baseline ECG and vital signs, laboratory values within normal limits (the lab tests include: complete blood count, electrolytes, liver function tests, kidney function tests, uric acid, cholesterol, iron, urinalysis, urine drug screen; all are conducted within 2 weeks prior to randomization).
* Women of Childbearing Potential (WCP) demonstrate a willingness to use contraception methods (other than birth control medications) to prevent pregnancy from time of consent to 30 days past last dose. **Note, birth control medications MAY BE used after completion of the inpatient hospital phase of the study (i.e. after discharge).
* Unremarkable past medical history.
* Ability to provide informed consent.
* Ability to undergo physical exercise (determined through a treadmill exercise test to ensure physical fitness of participants). Those who experience fatigue, dizziness or chest pain during the screening exercise test on the treadmill will be excluded.
* Ability to undergo neuropsychological test for attention, cognition, dexterity, etc.
* Willing to remain in the in-patient setting for the duration of the study.

Exclusion Criteria:

* Use of investigational drug within 4 weeks of study.
* Using tobacco.
* Acute illness or surgery within 4 weeks of study.
* Allergic to sulfonylurea-related drugs.
* Presence of pathological condition of any part of the body.
* Any medication within 2 weeks of the study, including oral contraceptives.
* Ingestion of alcohol or caffeine containing food or beverages within 48 hours of start of study.
* History of alcohol or drug abuse, cardiac arrhythmias, psychotropic agent use, immunosuppressive condition (i.e. HIV, AIDS, Cancer) or hepatitis.
* Donation of blood within 3 months or receiving blood products within 14 days.
* Recent body tattoo or piercing.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 7 days
  The primary objective of this study is to evaluate the safety of glyburide in healthy, non-diabetic volunteers while simulating strenuous activity to observe for any adverse events (i.e. hypoglycemia, dizziness, confusion, etc.). Neuropsychological testing, physical exams, vital signs, ECGs, cognitive assessments, and laboratory values (including serum glucose levels collected 4 x's per day and as needed) will be conducted throughout the 7 day in-patient study to assess for any adverse/serious adverse events.

SECONDARY OUTCOMES:
Cognitive impact | 7 days
  Determine the impact after 7 days of glyburide 1.5mg daily (with breakfast) in healthy volunteers who are able to participate in scheduled strenuous activities and adhere to a structured meal plan on cognitive performance using a computer program to test cognition before study drug administration and at the end of the study in addition to daily physical examinations which include mini mental status exams.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Bochicchio, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis Clinical Research Unit (CRU), St Louis, Missouri, United States